CLINICAL TRIAL: NCT04729764
Title: A Single-center, Randomized, Double-blind, Placebo-controlled and Single-center, Randomized, Open, Double-crossed Food Impact Trial to Evaluate the Safety, Tolerability, Pharmacokineticof GP681 Tablets in Healthy Subjects
Brief Title: Evaluation the Safety and Tolerance of GP681 Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: GP681101/CRC-C1933
Record Dates: First submitted 2020-08-27; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2020-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: According to the initial dose and maximum dose interval, it is designed as 5 dose groups (20mg, 40mg, 60mg, 80mg, 120mg), the initial dose group (20mg) has 8 subjects (including 2 placebo), and each of the others 10 subjects in the dose group (including 2 placebo), male and female.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This trial uses a double-blind technique, that is, neither the investigator nor the subject knows what kind of drug they are taking. The sponsor or its designated unit shall provide the trial drug and placebo to ensure that the placebo's shape, color, smell, taste, and weight are consistent with the trial drug, and the drug randomization and supply management system (RTSM) is used for drug randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- GP681 Tablet 20mg (Experimental): Two sentinel subjects were first enrolled in the trial (test drug: placebo=1:1). After the two sentinel subjects completed the 72h safety follow-up after the administration, it was judged that if there was no dose-limiting toxicity , Then start the trial of the remaining 6 subjects in the dose group (experimental drug: placebo = 5:1).
  Interventions: Drug: GP681 Tablet
- GP681 Tablet 40mg (Experimental): 10 subjects in 40mg group (including 2 placebo)
  Interventions: Drug: GP681 Tablet
- GP681 Tablet 60mg (Experimental): 10 subjects in 60mg group (including 2 placebo)
  Interventions: Drug: GP681 Tablet
- GP681 Tablet 80mg (Experimental): 10 subjects in 80mg group (including 2 placebo)
  Interventions: Drug: GP681 Tablet
- GP681 Tablet 120mg (Experimental): 10 subjects in 120mg group (including 2 placebo)
  Interventions: Drug: GP681 Tablet

INTERVENTIONS:
Drug: GP681 Tablet — Designed as 5 dose groups (20mg, 40mg, 60mg, 80mg, 120mg), the starting dose group (20mg) 8 subjects (including 2 placebo), each other 10 subjects (including Placebo (2 cases), male and female.

SUMMARY:
Influenza (influenza for short) is an acute respiratory infectious disease caused by influenza virus. The symptoms of the disease range from mild, moderate to severe, and severe cases require hospitalization and may die. According to estimates by the US Centers for Disease Control and Prevention in 2018, influenza causes approximately 290,000 to 640,000 deaths worldwide each year. Therefore, the prevention and treatment of influenza has become a serious public health problem.

DETAILED DESCRIPTION:
The GP681 in this test is a prodrug of a polymerase acidic protein (PA, Polymerase Acidic protein) inhibitor. Its metabolite GP1707D07 can selectively inhibit the cap-dependent endonuclease of influenza virus and prevent influenza virus replication. Mechanism of action against influenza virus. The results of previous non-clinical studies show that GP681 can effectively inhibit influenza virus replication, has good safety, and has antiviral activity 1,000 times that of oseltamivir phosphate. It also has good antiviral activity against oseltamivir resistant strains. And it is expected to have a longer half-life than oseltamivir phosphate. Therefore, it is expected that a new type of PA inhibitor can be developed to provide patients with influenza with a new mechanism of action, better efficacy, and higher compliance.

ELIGIBILITY:
Inclusion Criteria:

- 18-45 years old, male or female (the food impact test is limited to males); male ≥50 kg, female ≥45kg,BMI19-26; Fully understand the purpose and requirements of this trial, voluntarily participate in the clinical trial and sign a written informed consent form, and be able to complete the entire trial process according to the trial requirements.

Exclusion Criteria:

- history of allergies, allergic diseases or allergies to drugs in research; medical history of the central nervous system, cardiovascular system, digestive system, respiratory system, urinary system, blood system, metabolic disorders, etc. or other diseases that are not suitable for participating in clinical trials (such as mental illness history, etc.); donated blood or blood loss ≥ 400 mL within 3 months before enrollment;

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter | 12 days
  Peak concentration (Cmax)
ncidence of adverse events as a measure of safety and tolerability | 12 days
  Observed side effects and alteration in laboratory values.
area under the drug-time curve | 12 days
  area under the drug-time curve (AUC0-t, AUC0-∞)

CONTACTS AND LOCATIONS:
Overall Officials: liu yanmei, Principal Investigator — Shanghai Xuhui Central Hospital
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wu Q, Lv L, Yan S, Wang Y, Chen Q, Xu W, Liu Y, Wang W, Jia J, Yu C, Chen J, Liu Y. A first-in-human phase I study to evaluate the safety, tolerability, and pharmacokinetics of a novel anti-influenza agent suraxavir marboxil in healthy Chinese subjects. Antimicrob Agents Chemother. 2025 Nov 5;69(11):e0068525. doi: 10.1128/aac.00685-25. Epub 2025 Sep 30. PMID 41025645